CLINICAL TRIAL: NCT04188106
Title: Efficacy and Tolerability of Combination Varenicline With Hydroxyzine as a Potential Smoking Cessation Treatment
Acronym: HAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Principal Investigator, Jed Rose, President and CEO, Rose Research Center, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAVE
Record Dates: First submitted 2019-06-06; First posted 2019-12-05 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation; Stress; Sleep Disturbance; Nausea
MeSH Terms: conditions — Smoking Cessation; Parasomnias; Nausea | interventions — Varenicline; Hydroxyzine

STUDY DESIGN:
Intervention Model Description: Open-label, single group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hydroxyzine and Varenicline (Experimental): Participants enrolled in the study will take the FDA approved starter kit of varenicline for the first week of medication administration (0.5 mg nightly for days 1-3, then 0.5 mg twice daily for days 4-7). During the first week, participants will also receive hydroxyzine dosed in a similar manner, 50 mg nightly for the first 3 days, then twice daily, 25 mg in the morning and 50 mg at night. After the first week, participants will receive the FDA-approved dose of varenicline (1 mg twice daily) combined with hydroxyzine, 25 mg in the morning and 50 mg at nighttime. All medications will be dosed orally.
  Interventions: Drug: Varenicline Pill; Drug: Hydroxyzine Pill

INTERVENTIONS:
Drug: Varenicline Pill — FDA approved starter kit of varenicline (0.5 mg nightly for days 1-3, then 0.5 mg twice daily for days 4-7) followed by FDA-approved dose of varenicline (1 mg twice daily) for the remaining 11 weeks
  Other Names: Chantix
Drug: Hydroxyzine Pill — For the first week, participants will receive 50 mg nightly for the first 3 days, then twice daily, 25 mg in the morning and 50 mg at night for the remaining 12 weeks.

SUMMARY:
This open-label study will evaluate hydroxyzine, a first-generation antihistamine, combined with varenicline, to help smokers abstain from smoking during a 12-week trial period by diminishing the nausea, stress, anxiety, and sleep disturbances associated with the use of varenicline and with nicotine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the consent form and is able to read and understand the information provided in the consent form.
2. Is 19 to 65 years of age (inclusive) at screening.
3. Smokes at least 10 commercially available cigarettes per day for the last 12 months.
4. Has an expired air carbon monoxide reading of at least 10 ppm at screening.
5. Express a desire to quit smoking within the next 30 days at screening.
6. Willing and able to comply with the requirements of the study.
7. Participant owns a smart phone with text message and data capabilities.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. High blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
4. Body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2.
5. Coronary heart disease, structural cardiac disease, cardiac dysrhythmias, abnormal ECG (e.g. prolonged QTc), syncope, cardiac chest pain, or history of heart attack or heart failure.
6. Has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
7. Taking antidepressants, psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics) or medications that prolong QTc.
8. Positive urine drug test for cocaine, marijuana, opiates, amphetamines or methamphetamines.
9. Use of smokeless tobacco (chewing tobacco, snuff), cigars, pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of enrollment.
10. Pregnant or nursing (by self-report) or has a positive pregnancy test.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in both the Raleigh, NC and Charlotte, NC offices of Rose Research Center. Enrollment started on 17 June 2019 and ended on 16 September 2019.
Groups:
- Hydroxyzine and Varenicline: Participants enrolled in the study will take the FDA approved starter kit of varenicline for the first week of medication administration (0.5 mg nightly for days 1-3, then 0.5 mg twice daily for days 4-7). During the first week, participants will also receive hydroxyzine dosed in a similar manner, 50 mg nightly for the first 3 days, then twice daily, 25 mg in the morning and 50 mg at night. After the first week, participants will receive the FDA-approved dose of varenicline (1 mg twice daily) combined with hydroxyzine, 25 mg in the morning, and 50 mg at nighttime. All medications will be dosed orally.
Period: Overall Study
Arm/Group | Hydroxyzine and Varenicline
Started | 26
Completed | 20
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — Non-Compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxyzine and Varenicline
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.115 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in 10-item Perceived Stress Scale (PSS-10) Following Smoking Cessation (While Taking Arenicline and Hydroxyzine).
Description: Stress levels in the last 30 days will be measured using the 10-item Perceived Stress Scale (PSS-10). The PSS-10 uses a 5-point scale (0 - never, 1 = almost never, 2 = once in a while, 3 = often, 4 = very often). Total scores range from 0 to 40.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Time Frame: Weeks 1, 2, 4, 8, 12
Population: The number of participants changes based on dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydroxyzine and Varenicline
Number analyzed (Participants) | 24
score on a scale
  Change in PPS-10 from BL to Week 1 | -1.38 (2.37)
  Change in PPS-10 from BL to Week 2: number analyzed (Participants) | 23
  Change in PPS-10 from BL to Week 2 | -1.48 (3)
  Change in PPS-10 from BL to Week 4: number analyzed (Participants) | 22
  Change in PPS-10 from BL to Week 4 | -1.55 (2.65)
  Change in PPS-10 from BL to Week 8: number analyzed (Participants) | 22
  Change in PPS-10 from BL to Week 8 | -2.05 (3.58)
  Change in PPS-10 from BL to Week 12: number analyzed (Participants) | 20
  Change in PPS-10 from BL to Week 12 | -2.75 (3.43)

2. Primary Outcome: Changes in Anxiety Using the 6-item State-Trait Anxiety Inventory (STAI)
Description: Trait and state anxiety levels will be monitored for changes using the 6-item State-Trait Anxiety Inventory (STAI). All items are rated on a 4-point scale ("1-Almost Never" to "4-Almost Always"). The range of scores is from 6 to 24. Higher scores indicate greater anxiety.
Time Frame: Weeks 1, 2, 4, 8, 12
Population: The number of participants changes based on dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydroxyzine and Varenicline
Number analyzed (Participants) | 24
score on a scale
  Change in STAI from BL to Week 1 | -0.54 (2.67)
  Change in STAI from BL to Week 2: number analyzed (Participants) | 23
  Change in STAI from BL to Week 2 | -1.09 (3.79)
  Change in STAI from BL to Week 4: number analyzed (Participants) | 22
  Change in STAI from BL to Week 4 | -0.86 (4.54)
  Change in STAI from BL to Week 8: number analyzed (Participants) | 22
  Change in STAI from BL to Week 8 | -1.82 (3.35)
  Change in STAI from BL to Week 12: number analyzed (Participants) | 20
  Change in STAI from BL to Week 12 | -1.65 (3.59)

3. Primary Outcome: Changes in Depression Using the Patient Health Questionnaire (PHQ-9)
Description: Depression will be monitored for changes using the Patient Health Questionnaire (PHQ-9). The PHQ-9 uses a 4-point scale (Not at all = 0; Several days = 1;More than half the days = 2; Nearly every day = 3). The sum of the scores is calculated (Score range is 0 to 27):
  * 1-4 Minimal depression
  * 5-9 Mild depression
  * 10-14 Moderate depression
  * 15-19 Moderately severe depression
  * 20-27 Severe depression
Time Frame: Weeks 1, 2, 4, 8, 12
Population: The number of participants changes based on dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydroxyzine and Varenicline
Number analyzed (Participants) | 24
score on a scale
  Change in PHQ-9 from BL to Week 1 | -0.15 (1.12)
  Change in PHQ-9 from BL to Week 2: number analyzed (Participants) | 23
  Change in PHQ-9 from BL to Week 2 | 0.63 (2.16)
  Change in PHQ-9 from BL to Week 4: number analyzed (Participants) | 22
  Change in PHQ-9 from BL to Week 4 | 0.43 (2.95)
  Change in PHQ-9 from BL to Week 8: number analyzed (Participants) | 22
  Change in PHQ-9 from BL to Week 8 | -0.27 (2.07)
  Change in PHQ-9 from BL to Week 12: number analyzed (Participants) | 20
  Change in PHQ-9 from BL to Week 12 | -0.41 (1.87)

4. Secondary Outcome: Effects of Varenicline on Self-reported Smoking Reduction Prior to the Quit Date
Description: Previous research has shown that abstinence at the end of treatment is strongly predicted by the extent to which smokers spontaneously reduce ad libitum smoking in the initial weeks of pharmacotherapy that is initiated before the quit-smoking date.
  This measure will assess the extent of smoking reduction in participants during the initial seven days of treatment (prior to their planned quit date) - assessed via a self-report number of cigarettes per day. Data is recorded as a mean change.
Time Frame: 7 Days
Population: The participants are divided as to whether they were successful in quitting smoking combustible cigarettes.
Measure: Mean (Standard Deviation); unit: Cigs smoked per day
Groups:
- Hydroxyzine and Varenicline -- Successful in Quitting Smoking; Hydroxyzine and Varenicline -- Unsuccessful in Quitting Smoking: Participants enrolled in the study will take the FDA-approved starter kit of varenicline for the first week of medication administration (0.5 mg nightly for days 1-3, then 0.5 mg twice daily for days 4-7). During the first week, participants will also receive hydroxyzine dosed in a similar manner, 50 mg nightly for the first 3 days, then twice daily, 25 mg in the morning and 50 mg at night. After the first week, participants will receive the FDA-approved dose of varenicline (1 mg twice daily) combined with hydroxyzine, 25 mg in the morning, and 50 mg at nighttime. All medications will be dosed orally.
Arm/Group | Hydroxyzine and Varenicline -- Successful in Quitting Smoking | Hydroxyzine and Varenicline -- Unsuccessful in Quitting Smoking
Number analyzed (Participants) | 7 | 19
Cigs smoked per day | -9.14 (2.29) | -5.53 (6.80)

5. Secondary Outcome: Effects of Varenicline on Self-reported Smoking Reduction Prior to the Quit Date
Description: Previous research has shown that abstinence at the end of treatment is strongly predicted by the extent to which smokers spontaneously reduce ad libitum smoking in the initial weeks of pharmacotherapy that is initiated before the quit-smoking date.
  This measure will assess the extent of smoking reduction in participants during the initial seven days of treatment (prior to their planned quit date) - assessed via expired air carbon monoxide (CO). Data is recorded as a mean change.
Time Frame: 7 Days
Population: The participants are divided as to whether they were successful in quitting smoking combustible cigarettes.
Measure: Mean (Standard Deviation); unit: CO in ppm
Arm/Group | Hydroxyzine and Varenicline -- Successful in Quitting Smoking | Hydroxyzine and Varenicline -- Unsuccessful in Quitting Smoking
Number analyzed (Participants) | 7 | 19
CO in ppm | -11.00 (8.28) | -2.12 (10.02)

ADVERSE EVENTS:
Time Frame: Data were collected during the 12 week treatment period.
Arm/Group | Hydroxyzine and Varenicline
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 21/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyzine and Varenicline (N=26)
Hypersomnolence (Nervous system disorders) | 9 (11)
Nausea (Gastrointestinal disorders) | 10 (10)
Insomnia (Nervous system disorders) | 9 (9)
Mood Changes (Psychiatric disorders) | 7 (7)
Headache (Nervous system disorders) | 5 (5)
Elevated blood pressure (Cardiac disorders) | 4 (4)
Vivid dreams (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04188106/Prot_SAP_000.pdf